CLINICAL TRIAL: NCT02214589
Title: Non-pharmacological Interventions for Procedural Pain in Premature Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Danilyn Angeles, PhD, Professor, Loma Linda University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB5140027
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Prevention of Procedural Pain; Reduction of Procedural Pain; Biochemical Effects of Oral Dextrose
MeSH Terms: interventions — Glucose; Facilitated Tucking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral glucose and NNS (Active Comparator): Oral glucose and NNS
  Interventions: Other: Oral glucose and NNS
- Oral glucose and facilitated tucking and NNS (Active Comparator): Oral glucose, facilitated tucking and NNS
  Interventions: Other: Oral glucose, facilitated tucking, NNS
- Facilitated Tucking and NNS (Active Comparator): Facilitated tucking and NNS
  Interventions: Other: Facilitated tucking and NNS

INTERVENTIONS:
Other: Oral glucose, facilitated tucking, NNS
  Arms: Oral glucose and facilitated tucking and NNS
Other: Oral glucose and NNS
  Arms: Oral glucose and NNS
Other: Facilitated tucking and NNS
  Arms: Facilitated Tucking and NNS

SUMMARY:
A. Specific Aims Premature infants admitted to the neonatal intensive care unit (NICU) require up to several hundred procedures during their hospitalization. Many of these are tissue-damaging procedures (TDPs) known to cause pain [1]. Through funding from NINR, the investigators found that TDPs not only caused pain but also increased markers of ATP degradation and oxidative stress[2[. The TDP was tape removal, a commonly performed procedure in the NICU2.

Based on this finding, the investigators sought to determine if interventions that relieve pain also reduce biochemical markers of ATP degradation and oxidative stress. The investigators first examined the effect of oral sucrose, a commonly used intervention, when given before a heel lance. The investigators chose heel lance because it is the most predominant painful procedure in the NICU, as shown in 29 different clinical trials[3]. The investigators hypothesized that since oral sucrose is documented to significantly reduce pain scores, then administration of this analgesic will also decrease markers of ATP degradation and oxidative stress. However,the investigators observed the opposite effect. Although a single dose of oral sucrose reduced behavioral markers of pain, it significantly increased biochemical markers of ATP degradation (hypoxanthine, uric acid) and oxidative stress (allantoin) over time[4]. More importantly, the effect of oral sucrose on breakdown markers of ATP were enhanced and were significantly higher in neonates that were intubated or were receiving more than 30% FiO25. These findings lead to the question: If oral sucrose does not effectively reduce the biochemical effects of procedural pain, what intervention or groups of intervention will decrease both behavioral markers of procedural pain and reduce ATP utilization and oxidative stress in premature neonates? For this RO1 renewal, the investigators propose to test the individual and additive effects of two commonly used interventions for procedural pain. These interventions are (a) administration of 30% oral glucose and non-nutritive sucking (NNS) (b) facilitated tucking and NNS c) administration of 30% oral glucose, facilitated tucking and NNS. Administration of 30% oral glucose was documented to decreased procedural pain scores[6-9] without the potential adverse effects of fructose, a key ingredient of sucrose[10-11]. Facilitated tucking is the gentle positioning of preterm infants with arms and legs in a flexed, midline position close to the body, while either in a side-lying or prone position[12]. Because tachycardia often accompanies pain, a documented benefit of facilitated tucking is stabilization of heart rate and reduction of motor activity (flailing)[12-13]. Non-nutritive sucking refers to the provision of a weight-appropriate pacifier[14]. The painful procedure will be a clinically required heel lance, which refers to the puncture of a newborn's heel for blood glucose using a specially designed lancet. Our general hypothesis is that commonly used clinical interventions known to reduce procedural pain alter biochemical markers of ATP degradation, oxidative stress and cell injury.

Specific Aim 1 will determine whether (a) 30% oral glucose and NNS or (b) facilitated tucking and NNS or (c) 30% oral glucose with facilitated tucking and NNS will decrease procedural pain.

• Pain will be quantified using a validated pain scoring tool, the Premature Infant Pain Profile (PIPP). Individual and additive effect of interventions will be determined.

Specific Aim 2 will determine whether (a) 30% oral glucose and NNS or (b) facilitated tucking and NNS or (c) 30% oral glucose with facilitated tucking and NNS will decrease biochemical markers of ATP degradation, oxidative stress and oxidative cell injury.

* Products of ATP breakdown in plasma-hypoxanthine (Hx), xanthine (Xa), and uric acid (UA)-will be measured using high performance liquid chromatography.
* Oxidative stress will be quantified by measuring plasma levels of allantoin using mass spectrometry.
* Cell injury will be quantified by measuring plasma levels of F2 isoprostane using liquid-chromatography/mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects are premature infants between 28-36 weeks gestation, have an arterial or central catheter in place and have a clinically required heel lance.

Exclusion Criteria:

* Requirement for surgery
* Intraventricular hemorrhage (IVH) ≥ grade 3
* Neonates on medications such as morphine, fentanyl, versed, muscle relaxants, phenobarbital, or dilantin
* Renal injury (plasma creatinine > 1 mg/dl)
* Severe cyanotic heart disease or severe respiratory distress
* Chromosomal anomaly
* Facial anomaly

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Decreased pain score using the Premature Infant Pain Profile pain scoring tool | at time of heelstick
  A decrease in pain score will be quantified using the validated tool Premature Infant Pain Profile, which will be scored by a neonatologist blinded to group assignment.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States